CLINICAL TRIAL: NCT06836557
Title: A Multicenter, Open Label, 3-Month Safety Study with Tradipitant in Patients with Idiopathic or Diabetic Gastroparesis
Brief Title: Open Label Safety Study of Tradipitant in Idiopathic and Diabetic Gastroparesis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VLY-686-3304
Record Dates: First submitted 2024-04-01; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Gastroparesis; Diabetic Gastroparesis; Gastroparesis
Keywords: gastroparesis; idiopathic; diabetic; tradipitant; nausea; vomiting; stomach; motility; functional; NK-1 antagonist; neurokinin 1 receptor; substance p
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Tradipitant

INTERVENTIONS:
Drug: Tradipitant — BID

SUMMARY:
This is a multicenter, open label, 3-month safety study with tradipitant in patients with idiopathic and diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastroparesis
* Demonstrated delayed gastric emptying
* Presence of moderate to severe nausea
* Body Mass Index (BMI) of ≥18 and ≤40 kg/m2

Exclusion Criteria:

* Another active disorder or treatment which could explain or contribute to symptoms of gastroparesis
* A positive test for drugs of abuse at the screening or evaluation visits
* Pregnancy or nursing
* Evidence of uncontrolled blood glucose (including HbA1C >11% at screening or metabolic crisis in past 60 days)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), including suicidal ideation or behavior as measured by the C-SSRS | 12 weeks
  AEs will be coded using the MedDRA coding dictionary. An AE is defined as any untoward medical occurrence in a clinical investigation subject that does not necessarily have causal relationship with treatment. AEs will further be categorized by severity, relationship to study medication, and action taken. All AEs will be presented in data listings for subjects.
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a semi-structured clinical interview designed to systematically assess and track suicidal adverse events (behavior and ideation) throughout different settings including clinical trials. Results from the C-SSRS will be listed for each subject. These data will also be summarized for all subjects for suicidal ideation events, suicidal behaviors, and completed suicides.
Number of participants with changes in vital signs identified as Clinically Notable Abnormal values | 12 weeks
  Vital sign measurements include oral temperature (C), respiratory rate, semi-supine blood pressure (systolic and diastolic) (mmHg) and semi-supine heart rate (bpm). Criteria for identifying vital signs as Potentially Clinically Notable Abnormalities are based on the Guidelines for the Division of Neuropharmacological Drug Products. Data from vital signs will be listed, clinically notable values will be flagged, and other information collected will be listed. Data will also be summarized using mean change from first study visit and proportion of subjects with values outside the normal range, and values that were clinically notable.
Number of participants with abnormal and potentially Clinically Notable Abnormal Electrocardiogram Intervals and Heart Rate | 12 weeks
  Variables include PR (ms), QRS (ms), QTc (ms), and Heart Rate (bpm). Note: ms = millisecond; bpm = beats per minute
Number of participants with Clinically Notable Abnormal laboratory values | 12 weeks
  Laboratory data will be summarized by presenting the proportions of patients with clinically notable abnormalities as follows: shift tables, first study visit to most extreme post-treatment value, using normal ranges; summary statistics of raw data and change from first study visit values (means, medians, standard deviations, ranges). Criteria for identifying laboratory values as Potentially Clinically Notable Abnormalities are based on the FDA's Guidelines for the Division of Neuropharmacological Drug Products.

SECONDARY OUTCOMES:
To evaluate the efficacy of tradipitant in reducing individual symptoms associated with gastroparesis | 12 weeks
  Efficacy is assessed by the Gastroparesis Core Symptom Daily Diary (GCSDD). The GCSDD is a daily symptom diary asking patients to rate their nausea on a Likert scale from 0-5 (0=none, 5= very severe). Other symptoms include vomiting, postprandial fullness, early satiety, and abdominal pain.
To evaluate the efficacy of tradipitant in global improvement | 12 weeks
  Efficacy is assessed by the Clinical Global Impression - Severity (CGI-S). The CGI-S is a clinician reported outcome that measures the clinician's view of the patient's global functioning prior to and after initiating treatment. Symptom severity is measured on a 7 point scale including "1=normal, not at all ill" and "7=among the most extremely ill patients."

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (3):
- Belgium (2):
  - Vanda Investigational Site, Leuven
  - Vanda Investigational Site, Liège
- Vanda Investigational Site, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No